CLINICAL TRIAL: NCT02484703
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group 26-Week Dose-Investigating Study to Explore the Pharmacokinetics, Pharmacodynamic Effects, Efficacy, Safety and Tolerability of RO5186582 in Children With Down Syndrome Aged 6-11 Years
Brief Title: A Study of RO5186582 in Down Syndrome Among Children 6 to 11 Years of Age
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to data from another study showing no efficacy. There were no safety issues of concern.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WP28760
Record Dates: First submitted 2015-06-16; First posted 2015-06-30 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Placebo (Placebo Comparator): Participants will receive matching placebo by mouth (PO) twice daily (BID) for up to 26 weeks.
  Interventions: Drug: Placebo
- RO5186582 120 mg BID (Experimental): Participants will receive RO5186582 at a dosage of 120 milligrams (mg) PO BID for up to 26 weeks.
  Interventions: Drug: RO5186582
- RO5186582 40 mg BID (Experimental): Participants will receive RO5186582 at a dosage of 40 mg PO BID for up to 26 weeks.
  Interventions: Drug: RO5186582
- RO5186582 60 mg BID (Experimental): Participants will receive RO5186582 at a dosage of 60 mg PO BID for up to 26 weeks.
  Interventions: Drug: RO5186582

INTERVENTIONS:
Drug: Placebo — Participants will receive matching placebo PO BID. Study medication will first be administered on Day 1, and only the morning dose will be given on the last day of treatment (Week 26).
  Arms: Placebo
Drug: RO5186582 — Participants will receive 1 of 3 dosages of RO5186582 PO BID, including 40 mg, 60 mg, or 120 mg. Study medication will first be administered on Day 1, and only the morning dose will be given on the last day of treatment (Week 26).
  Arms: RO5186582 120 mg BID; RO5186582 40 mg BID; RO5186582 60 mg BID

SUMMARY:
This study will evaluate the safety, tolerability, efficacy, and pharmacokinetic and pharmacodynamic activity of 3 different dosages of RO5186582 compared with placebo. A total of approximately 46 participants will be enrolled, in order to have at least 32 evaluable, and will be randomly assigned to 1 of 4 treatments in a 1:1:1:1 ratio, with 9 children per treatment arm. The target ratio between 6-8 years and 9-11 years age groups is approximately 1:1 in each treatment arm, with a minimum of 3 children per age group in each treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Down syndrome, except for mosaic Down syndrome
* Available parent or caregiver to attend clinic visits and provide information about the participant's behavior and symptoms

Exclusion Criteria:

* Any primary psychiatric comorbid disorder
* History of infantile spasms, West syndrome, Lennox-Gastaut syndrome, early infantile epileptic encephalopathy, treatment-refractory epilepsy with cognitive/developmental regression, severe head trauma, or central nervous system (CNS) infection
* Seizure event of any type within 12 months prior to Screening or relevant changes in anti-epileptic drugs 6 weeks prior to enrollment
* Significant sleep disruption
* Significant gastrointestinal, renal, hepatic, endocrine, or cardiovascular disease
* New-onset or ongoing hematologic/oncologic disorder
* Severe lactose intolerance
* Participation in another clinical study within 1 month or 6 half-lives prior to first dose, or any extent of participation in Study BP29589 (NCT02451657)

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2015-10-28 (Actual); Primary Completion 2016-08-03 (Actual); Study Completion 2016-08-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) | Baseline up to Week 6
Percentage of Participants With Epileptiform Abnormalities as Assessed Using Electroencephalogram (EEG) Analysis | Baseline up to Week 6
Percentage of Participants by Suicidality Classification as Assessed Using an Adapted Form of the Columbia Classification Algorithm for Suicide Assessment (C-CASA) | Baseline up to Week 6
Anxiety, Depression, and Mood Scale (ADAMS) Score | Baseline up to Week 6
Hyperactivity and Impulsivity as Assessed by the Short Version of Conners Third Edition Parent Short-Form (Conners-3) Score | Baseline up to Week 6
Sleep Disturbances as Assessed by the Children's Sleep Habits Questionnaire (CSHQ) Score | Baseline up to Week 6
Gamma Power at Posterior Electrodes as Assessed Using EEG Analysis | Baseline up to Week 6
Theta Power at Posterior Electrodes as Assessed Using EEG Analysis | Baseline up to Week 6
Cognition as Assessed by the Children's Memory Scale (CMS) Subtests Score | Baseline up to Week 6

SECONDARY OUTCOMES:
Percentage of Participants With AEs | Baseline up to Week 26
Percentage of Participants With Epileptiform Abnormalities as Assessed Using EEG Analysis | Baseline up to Week 26
Percentage of Participants by Suicidality Classification as Assessed Using an Adapted Form of the C-CASA | Baseline up to Week 26
ADAMS Score | Baseline up to Week 26
Hyperactivity and Impulsivity as Assessed by the Short Version of Conners-3 Score | Baseline up to Week 26
Sleep Disturbances as Assessed by the CSHQ Score | Baseline up to Week 26
Gamma Power at Posterior Electrodes as Assessed Using EEG Analysis | Baseline up to Week 26
Theta Power at Posterior Electrodes as Assessed Using EEG Analysis | Baseline up to Week 26
Cognition as Assessed by the CMS Subtests Score | Baseline up to Week 26
Adaptive Behavior as Assessed by the Vineland Adaptive Behavior Scales-II (VABS-II) Score | Baseline up to Week 26
Clinical Global Impression-Improvement (CGI-I) Scale Score | Baseline up to Week 26
Daily Functional Memory as Assessed by the Observer Memory Questionnaire-Parent Form (OMQ-PF) Score | Baseline up to Week 26
Intellectual Quotient (IQ) as Assessed by the Leiter 3 | Baseline up to Week 26
Plasma Concentration of RO5186582 | Predose (2 predose samples separated by at least 1 hour) at Weeks 2 and 6; and predose or postdose (as convenient) during Weeks 10, 17, and 26

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- United States (9):
  - Southwest Autism Research & Resource Center, Phoenix, Arizona
  - Emory University School of Medicine; Department of Human Genetics & Pediatrics, Decatur, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Massachusette General Hospital; Medical Genetics, Boston, Massachusetts
  - Boston Children's Hospital, Department of Neurology, Boston, Massachusetts
  - Duke Clin Rsch Institute, Durham, North Carolina
  - UPMC Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin